CLINICAL TRIAL: NCT02284139
Title: Pilot Trial of Epidermal Growth Factor (EGF) Ointment for the Patients With Epidermal Growth Factor Receptor (EGFR) Inhibitor Related Skin Side Effects
Brief Title: Pilot Trial of EGF Ointment for the Patients With EGFR-i Related Skin Side Effects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, Sung Yong Oh, Department of Internal Medicine, Dong-A University Hospital, Dong-A University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAUH-14-211
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Non-small Cell Lung Cancer; Pancreatic Cancer; Colorectal Cancer
Keywords: EGF ointment; EGFR inhibitor; Skin side effect
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo ointment dose not contain EGF.
  Interventions: Drug: Arm Placebos
- Arm EGF ointment 1ppm (Active Comparator): Arm EGF ointment 1ppm will be treated with EGF ointment of 1 ppm concentration
  Interventions: Drug: Arm EGF ointment 1ppm
- Arm EGF ointment 20ppm (Active Comparator): Arm EGF ointment 20ppm will be treated with EGF ointment of 20 ppm concentration
  Interventions: Drug: Arm EGF ointment 20 ppm

INTERVENTIONS:
Drug: Arm EGF ointment 1ppm — EGF Ointment 1ppm evenly apply to skin lesion every 12 hr/ day
  Other Names: Saesal yeongo 1 (EGF ointment 1ppm)
  Arms: Arm EGF ointment 1ppm
Drug: Arm EGF ointment 20 ppm — EGF Ointment 20 evenly apply to skin lesion every 12 hr/ day
  Other Names: Saesal yeongo 20 (EGF ointment 20 ppm)
  Arms: Arm EGF ointment 20ppm
Drug: Arm Placebos — EGF Ointment 0ppm evenly apply to skin lesion every 12 hr/ day
  Other Names: Saesal yeongo 0 (EGF ointment 0 ppm)
  Arms: Placebo

SUMMARY:
The efficacy of the epidermal growth factor receptor (EGFR) inhibitors have been demonstrated in patients with non-small cell lung cancer (NSCLC), pancreatic cancer (PC) and colorectal cancer (CRC). Dermatological reactions can cause significant physical and psycho-social discomfort to patients. In the present study, the investigators evaluated the effect of epidermal growth factor (EGF) ointment on EGFR inhibitor-related skin side effects (ERSEs).

DETAILED DESCRIPTION:
The current study includes patients diagnosed with advanced NSCLC or PC or CRC, with pathological confirmation. The inclusion criteria were NSCLC treated with erlotinib alone and PC treated with gemcitabine and erlotinib combination chemotherapy and CRC treated with cetuximab and5-Fluorouracil (5-FU)+Irinotecan+leucovorin(LV) (FOLFIRI), 5-FU+Oxaliplatin+LV (FOLFOX) and sufficient liver, kidney, and bone marrow function to undergo treatment. All the patients had Grade ≥2 ERSEs according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) v. 4.03.

The patients will be randomized 3 groups; Placebo group, Arm 1, and Arm 2. Arm 1 will be treated with 1ppm concentration EGF ointment. Arm 2 will be treated with 20ppm concentration EGF ointment. And placebo group will be treated with 0ppm concentration EGF ointment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: older than 20
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 -2
3. Histologically confirmed lung cancer, pancreatic cancer, or colon cancer
4. Patients take EGFR inhibitor following the reason

   * EGFR mutation (+) NSCLC - adenocarcinoma for 1st line treatment
   * NSCLC - for ≥ 2nd line treatment
   * Pancreatic cancer - adenocarcinoma for 1st line treatment with Gemcitabine
   * Colon cancer - adenocarcinoma 1st line treatment with Irinotecan (FOLFIRI)
5. Patients who have EGFR inhibitor related skin side effects (ERSE) Gr≥2 (NCICTC V4.0)
6. A patient with the willingness to comply with the study protocol during the study period and capable of complying with it
7. A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages

Exclusion Criteria:

1. A patient with previous active or passive immunotherapy
2. A pregnant or lactating patient
3. A patient of childbearing potential without being tested for pregnancy at baseline for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential.)
4. A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications
5. A patient with history of dermatologic care (except transient urticaria) within 4 weeks
6. A patient with clinically significant (i.e. active) heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmias, etc) or myocardial infarction within past 12 months
7. A patient with interstitial pneumonia or diffused symptomatic fibrosis of the lungs.
8. Organ allogenic transplantation requiring immunosuppressive therapy. Any waiver of these inclusion and exclusion criteria must be approved by the investigator and the sponsor on a case-by case basis prior to enrolling the subject
9. Known allergies, hypersensitivity, or intolerance to study drugs, chemotherapy drugs using this clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To estimate the response rate of EGF ointment | 1 year
  The effectiveness of the EGF ointment was defined as follows:
  1. Grade 2, 3, or 4 ERSEs downgraded to ≤Grade 1 or
  2. Grade 3 or 4 ERSEs downgraded to Grade 2 and persisting for at least two weeks.

SECONDARY OUTCOMES:
Quality of Life | 1 year
  To evaluate the patients' Quality of Life (QoL) by Skin evaluation method (SKINDEX-16)

CONTACTS AND LOCATIONS:
Overall Officials: SUNG YONG OH, M.D., Principal Investigator — Dong-A University Hospital
Locations (1):
- Sung Yong Oh, Busan, South Korea

REFERENCES:
- [Derived] Kim YS, Ji JH, Oh SY, Lee S, Huh SJ, Lee JH, Song KH, Son CH, Roh MS, Lee GW, Lee J, Kim ST, Kim CK, Jang JS, Hwang IG, Ahn HK, Park LC, Oh SY, Kim SG, Lee SC, Lim DH, Lee SI, Kang JH. A Randomized Controlled Trial of Epidermal Growth Factor Ointment for Treating Epidermal Growth Factor Receptor Inhibitor-Induced Skin Toxicities. Oncologist. 2020 Jan;25(1):e186-e193. doi: 10.1634/theoncologist.2019-0221. Epub 2019 Sep 6. PMID 31492766